CLINICAL TRIAL: NCT07054710
Title: Eurofins CRL Cosmetics, Inc. / "A Clinical Study to Evaluate the Efficacy and Consumer Perception of a Cosmetic Device and Obtain Images"
Brief Title: Evaluation of the Efficacy of a Cosmetic Light Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Therabody, Inc. (Industry)
Collaborators: Eurofins CRL Cosmetics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECRLNJ2025-0269 BI
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Fine Lines; Contour; Sagging Skin; Dark Spots; Wrinkles; Firmness; Skin Tone; Radiance/Luminosity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Daily LED and Vibration Use (Experimental): Participants will use the device once daily for 12-15 minutes for 12-weeks. The device delivers LED (red light, red+infrared, and blue light) and vibration to the eye and scalp area.
  Interventions: Device: LED Light Treatment; Device: Vibration Only

INTERVENTIONS:
Device: LED Light Treatment — The device will guide participants through a treatment that cycles through Red (4 minutes), Red + Infrared (4 minutes), and Blue (4 minutes) LED therapy in combination with vibration therapy, for a 12-minute treatment. Participants will be asked to use the device Monday through Saturday, on a clean face, as part of their evening routine.
Device: Vibration Only — On each Sunday of the 12-week program, participants will be asked to complete a 15-minute vibration-only treatment session as part of their evening routine.

SUMMARY:
The present study evaluated facial skin health over a 12-week period using an at-home device that provides 12 minutes of LED light and vibration once daily, six days a week. The primary question it seeks to answer is whether daily use of the TheraFace Mask Glo alters facial skin characteristics. Secondary aims include collecting clinical images, professional photographs, and consumer perceptions of the device.

Participants between the ages of 39-64 with various skin types were enrolled for participation. Participants visited the clinic three times for collection of outcome metrics at baseline, 8 weeks, and 12 weeks. Participants also came to the lab at 4 weeks for a compliance check. Measurements included: expert clinical grading, digital imaging, subjective assessment of skin, and clinical grade-images.

DETAILED DESCRIPTION:
Light-emitting diode (LED) light therapy has recently gained popularity as a treatment for various skin conditions, such as fine lines, wrinkles, and age spots. LED treatments that use different wavelengths, like red, blue, and infrared, have been adapted into at-home devices to make these treatments more affordable and accessible for consumers. The main objective of this study is to assess the impact of an at-home LED treatment on skin health over 12 weeks. Participants completed a 12-minute LED + vibration treatment using the Therabody TheraFace Mask Glo at home six days a week for 12 weeks. The seventh day of each week involved a 15-minute vibration-only treatment. Outcome measures included measures of skin health in the face.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female or male (approximately 90% female and 10% male)
* Subject is between the ages of 35-65
* Male subjects agree to remove all facial hair 24-48 hours prior to each visit and remain clean shaven daily throughout the study
* Subject is of any Fitzpatrick (at least one of each, to be recorded)
* Subject is of any of the following (Caucasian, African American, Asian, Hispanic) (at least one of each, to be recorded)
* Subject has Self-Perceived Sensitive skin or Self-Perceived Non-Sensitive skin (approximately 50% sensitive and 50% non-sensitive)
* Subject has the following on face (mild or greater):

Fine lines, ≥3 on 10-point scale Wrinkles, ≥3 on 10-point scale Dull skin, ≥3 on 10-point scale Sagging, ≥3 on 10-point scale Uneven skin tone Roughness/texture At least one dark spot

* Subject agrees to return all used and unused test materials at the end of the study
* Subjects will use their regular SPF product or will use an SPF product provided by the Sponsor (if they do not have an SPF product) and practice sun safe practices for the duration of the study (Hat, sunglasses, etc.)
* Subject agrees not to introduce any new cosmetic or toiletry products during the study other than the products provided in this study
* Subject is willing to use a cosmetic device on their face
* Subject is dependable and able to follow directions as outlined in the protocol and anticipates being available for all study visits
* Subject is willing to participate in all study evaluations
* Subject is in generally good health and has a current Panelist Profile Form on file at ECRL
* Subject agrees to sign a Photography Release Form, providing consent for the capture of digital images for use in relation to this clinical study
* Subject has completed a HIPAA Authorization Form in conformance with 45 CFR Parts 160 and 164
* Subject understands and has signed an Informed Consent Form in conformance with 21 CFR Part 50: "Protection of Human Subjects."

Exclusion Criteria

* Female subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control
* Subject has been part of a clinical test for a LED device, microcurrent device or other facial device within the last 6 months
* Subject has eye sensitivity to light that may interfere with the use/application of the test product
* Subject has received treatment with sympathomimetics, antihistamines, vasoconstrictors, non-steroidal anti-inflammatory agents, and/or systemic or topical corticosteroids within one week prior to initiation of the study
* Subject has a history of acute or chronic dermatologic, medical, and/or physical conditions which would, in the opinion of the Principal Investigator, preclude application of the test material and/or could influence the outcome of the study
* Subject has a history of atopic eczema, psoriasis, or onychomycosis
* Subject chronically uses substances such as alcohol, tobacco, recreational drugs, etc.
* Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study
* Subject exhibits any facial tattoos/tattooed cosmetics, eyelash extensions, rashes, scratches, scars, or burn marks on the test site (face) which may interfere with the study
* Subject has known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs
* Subject is unable to communicate or cooperate with the Principal Investigator, language problems, etc.
* Subject is on another study utilizing the same test sites (Face)
* Subject is an employee of testing firms/laboratories, cosmetic or raw goods manufacturers or suppliers
* Subject has any planned medical or cosmetic procedures planned during the course of the study that, at the discretion of the Principal Investigator, may interfere with the study
* Subject has a history of skin cancer, or is currently undergoing treatment for active cancer of any kind
* Subject has diabetes.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Overall skin health appearance | 12-weeks
  Expert clinical grading, VISIA-CR imaging and participant perceptions will be used in conjunction to measure a variety of skin health appearance measures including: fine lines, wrinkles (including wrinkle depth), skin tone evenness, skin texture, firmness, contour, sagging skin, skin radiance and luminosity, skin texture and smoothness, and dark spot/aging spot appearance. The VISIA-CR is a clinical facial imaging system used to analyze skin conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins CRL Cosmetics, Inc, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No